CLINICAL TRIAL: NCT04170062
Title: Oxygen Savings With Administered Oxygen and High Flow Ambient Air At Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American College of Chest Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00206318
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pulmonary Fibrosis; Hypoxemia; Dyspnea; Oxygen Inhalation Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pulmonary Fibrosis; Hypoxia; Dyspnea | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Order of treatments tested will be randomized and only known to the person administering the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Baseline followed by intervention 1a (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 15 L/min, 20 L/min, 25 L/min) and then Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 15 L/min, 20 L/min, 25 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 1b (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 15 L/min, 25 L/min, 20 L/min) and then Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 15 L/min, 25 L/min, 20 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 1c (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 20 L/min, 15 L/min, 25 L/min) and then Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 20 L/min, 15 L/min, 25 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 1d (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 20 L/min, 25 L/min, 15 L/min) and then Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 20 L/min, 25 L/min, 15 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 1e (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 25 L/min, 15 L/min, 20 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 25 L/min, 15 L/min, 20 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 1f (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 25 L/min, 20 L/min, 15 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 25 L/min, 20 L/min, 15 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2a (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 15 L/min, 20 L/min, 25 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 15 L/min, 20 L/min, 25 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2b (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 15 L/min, 25 L/min, 20 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 15 L/min, 25 L/min, 20 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2c (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen order of high-flow air flow rate: 20 L/min, 15 L/min, 25 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 20 L/min, 15 L/min, 25 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2d (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 20 L/min, 25 L/min, 15 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 20 L/min, 25 L/min, 15 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2e (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 25 L/min, 15 L/min, 20 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 25 L/min, 15 L/min, 20 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy
- Baseline followed by intervention 2f (Experimental): Subjects perform baseline titration with oxygen only first. Subjects are then titrated with six different delivery methods. The subjects will be first delivered Out-of-Phase pulsed high-flow air and oxygen (order of high-flow air flow rate: 25 L/min, 20 L/min, 15 L/min) and then Continuous high-flow air with pulsed oxygen (order of high-flow air flow rate: 25 L/min, 20 L/min, 15 L/min).
  Interventions: Device: Nasal Delivery of High-Flow Air and Oxygen Therapy; Device: Nasal Delivery of Oxygen Therapy

INTERVENTIONS:
Device: Nasal Delivery of High-Flow Air and Oxygen Therapy — They will receive high-flow air and oxygen via a dual lumen nasal cannula at rest. Participants will be administered the high-flow air and then titrated with oxygen from 0 L/min until they reach and maintain a SpO2 level of 95% for 30 seconds. They will then remain on this setting for 3 additional minutes with continuous monitoring of SpO2 levels.
Device: Nasal Delivery of Oxygen Therapy — They will receive oxygen via a dual lumen nasal cannula at rest. Participants will be titrated with oxygen from 0 L/min until they reach and maintain a SpO2 level of 95% for 30 seconds. They will then remain on this setting for 3 additional minutes with continuous monitoring of SpO2 levels.

SUMMARY:
This study is meant to compare the amount of oxygen required for hypoxemia relief between current standard of care (oxygen only) and oxygen with the addition of high flow air for Chronic Obstructive Pulmonary Disease (COPD), Interstitial Lung Disease (ILD), and Pulmonary Hypertension (PH) patients during rest. Subjects will be titrated from 0 L/min until they maintain 95% SpO2 for each of the following delivery methods:

1. Pulses of pure oxygen (control)
2. Constant high flow air with pulses of pure oxygen
3. Out of phase pulses of high flow air and pure oxygen

DETAILED DESCRIPTION:
Each participant will require (1) visit, which will last approximately 4-5 hours.

At start of visit:

1. Vitals are taken (temperature, heart rate, SpO2, respiration rate, blood pressure, Borg dyspnea score, Mmrc score) while participant is seated and using their normal oxygen prescription.
2. Patient will remain seated during the following procedure with SpO2 and heart rate continuously being monitored.

Pulsed Oxygen Control at Rest:

1. Participant's oxygen will be turned off for 10 minutes as a washout period.
2. Using the oxygen tank with the pulse regulator, the participant will be titrated to a pulse rate that maintains their SpO2 at an average of 95%.

   a. Increasing volumes of oxygen in 1 L(liter)/min increments every thirty seconds until an average of 95% SpO2 is maintained for 30 seconds.
3. Once the participant is titrated to the correct amount of oxygen, they will remain on the oxygen for an additional 3 minutes
4. Final oxygen flow rate, SpO2, Heart Rate, and Borg Dyspnea Score will be recorded in the last minute of the test.

   Mixed Continuous Air/Oxygen Efficacy at Rest:
5. Participant's oxygen will be turned off for 10 minutes as a washout period.
6. The participant will be delivered pulsed oxygen and high flow ambient air using the oxygen tank with the pulse regulator and Vapotherm setup, the participant will be titrated to a pulse rate that maintains their SpO2 at an average of 95%.

   1. High flow ambient air will be set to 15 L/min
   2. Increasing volumes of oxygen from in 1 L/min increments every thirty seconds until an average of 95% SpO2 is maintained for 30 seconds.
7. Once the participant is titrated the correct amount of oxygen, they will remain on the oxygen for an additional 3 minutes.
8. Final oxygen flow rate, SpO2, Heart Rate, and Borg Dyspnea Score will be recorded in the last minute of the test.
9. Steps 5-8 are then repeated two more times for pulsed oxygen plus continuous flow ambient air at flow rates of 20 and 25 L/min.

   Mixed Pulsed Air/Oxygen Efficacy at Rest:
10. Participant's oxygen will be turned off for 10 minutes as a washout period
11. The participant will be delivered the out-of-phase pulsed oxygen and high flow ambient air using the oxygen tank with the pulse regulator and Vapotherm setup, the participant will be titrated to a pulse rate that maintains their SpO2 at an average of 95%

    1. High flow ambient air will be set to 15 L/min
    2. Increasing volumes of oxygen from in 1L/min increments every thirty seconds until an average of 95% SpO2 is maintained for 30 seconds.
12. Once the participant is titrated the correct amount of oxygen, they will remain on the oxygen for an additional 3 minutes
13. Final oxygen flow rate, SpO2, Heart Rate, and Borg Dyspnea Score will be recorded in the last minute of the test.
14. Steps 10-13 are then repeated two more times for out-of phase pulsed oxygen plus pulsed high flow ambient air at flow rates of 20 and 25 L/min.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged greater or equal to 30 years old
* Require Long Term Oxygen Therapy between 1 L/min and 4 L/min while at rest
* Have a peripheral blood saturation level above 80% with room air while seated
* Tolerate breathing while seated in room air
* Diagnosed with one of the following respiratory diseases: COPD (40% < Forced Expiratory Volume (FEV1) < 80% confirmed from pulmonary function test (PFT) within the last year), ILD (Confirmed with radiographic imaging), PH (Confirmed with radiographic imaging)
* Normal heart rate and blood pressure (Resting Heart Rate <120 bpm, Systolic BP <180 mmHg, Diastolic BP <100mmHg)
* PFT taken in the last three months

Exclusion Criteria:

* Pregnancy or lactation
* Exacerbation that has resolved within the past 28 days
* Treatment with another investigational drug or other intervention within three months
* Has any of the following: unstable angina, recent revascularization, recent history of cerebrovascular accident

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Effectiveness of partial replacement of concentrated oxygen by high flow ambient air for Long Term Oxygen Therapy | up to 20 minutes
  This will be assessed using the difference between the oxygen delivery systems (pure oxygen and mixed high-flow air with oxygen) in the L/min flow of oxygen required for a participant to reach steady state at greater than or equal to 95% pulse oxygenation.

SECONDARY OUTCOMES:
Dyspnea relief achieved with of partial replacement of concentrated oxygen by high flow ambient air for Long Term Oxygen Therapy | Approximately 15 minutes
  This will be assessed using the difference in relative dyspnea score evaluated with the Borg Dyspnea scale at the end of each delivery method. The Borg scale ranges from 0-10. Min: 0 (No dyspnea), Max: 10 (Very,Very Severe dyspnea).

CONTACTS AND LOCATIONS:
Overall Officials: Sonye Danoff, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital Bayview Asthma and Allergy Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No